CLINICAL TRIAL: NCT01406704
Title: Effects of Rosiglitazone and Alpha-lipoic Acid on the Patients With Pathologically Proved NASH (Non-alcoholic Steato-hepatitis)
Brief Title: Effects of Rosiglitazone and Alpha-lipoic Acid on the Patients With Pathologically Proved NASH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: because of withdrawal of Avandia sale due to its risks outweigh its benefits
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Kun Ho Yoon/principal investigator, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KCMC-04-14
Record Dates: First submitted 2011-07-27; First posted 2011-08-01 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2004-01

CONDITIONS: NASH (Non-alcoholic Steato-hepatitis)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Rosiglitazone; Thioctic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention)
- Rosiglitazone (Experimental): Rosiglitazone (8 mg/day)
  Interventions: Drug: Rosiglitazone
- alpha-lipoic acid (Experimental): alpha-lipoic acid (1800 mg/day)
  Interventions: Drug: alpha-lipoic acid
- Rosiglitazone/alpha-lipoic acid (Experimental): combination of Rosiglitazone (8 mg/day) and alpha-lipoic acid (1800 mg/day)
  Interventions: Drug: Rosiglitazone/alpha-lipoic acid

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone (8 mg/day)
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: alpha-lipoic acid — alpha-lipoic acid (1800 mg/day)
  Other Names: Thioctic acid
  Arms: alpha-lipoic acid
Drug: Rosiglitazone/alpha-lipoic acid — combination of Rosiglitazone (8 mg/day) and Thioctic acid (1800 mg/day)
  Other Names: Avandia/Thioctic acid
  Arms: Rosiglitazone/alpha-lipoic acid

SUMMARY:
This study is to evaluate the effects of Rosiglitazone, insulin sensitizer and alpha-lipoic acid, antioxidant on patients with pathologically proved NASH (non-alcoholic steato-hepatitis).

DETAILED DESCRIPTION:
Duration: 24 week-intervention Study Group: Four arms

* Control: no intervention
* Rosiglitazone: rosiglitazone (8 mg/day)
* alpha-lipoic acid: alpha-lipoic acid (1800 mg/day)
* Rosiglitazone/alpha-lipoic acid: combination of rosiglitazone (8 mg/day) and alpha-lipoic acid (1800 mg/day)

ELIGIBILITY:
Inclusion Criteria:

* the patients with pathologically proved NASH (non-alcoholic steato-hepatitis)

Exclusion Criteria:

* alcohol consumption > 20g/day
* viral hepatitis B and C
* autoimmune hepatitis
* Wilson's disease
* hemochromatosis
* alpha-1 antitrypsin deficiency
* breast-feeding or pregnant females
* subjects planning to become pregnant
* severe comorbid medical conditions (such as severe cardiac, pulmonary, renal or psychological problems)
* those not consenting for the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Histological evaluation | 24 weeks
  NASH Histological scoring system

SECONDARY OUTCOMES:
Biomechanical measurement | 24 weeks
  liver function test, insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Kun Ho Yoon, Principal Investigator — Seoul St. Mary's Hospital